CLINICAL TRIAL: NCT04890197
Title: The Effects of Tahini Consumption on Radiotherapy Induced Dermatitis in Breast Cancer - A Pilot Study
Brief Title: Tahini and Dermatitis in Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, professor, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1400
Record Dates: First submitted 2021-05-05; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tahini (Active Comparator): 48 gr per day
  Interventions: Dietary Supplement: tahini
- control (Placebo Comparator): no intervention
  Interventions: Other: control

INTERVENTIONS:
Dietary Supplement: tahini — 48 grams tahini
  Arms: tahini
Other: control — no intervention
  Arms: control

SUMMARY:
This study aimed to investigate the effect of tahini on acute radiation dermatitis in breast cancer (BC) patients undergoing radiotherapy (RT).

50 eligible BC patients will randomly assign to consume tahini 48 gr per day during and 1 week after RT or with no intervention (control group). The radiation dermatitis will be assessed weekly according to the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/EORTC) scales.

ELIGIBILITY:
Inclusion Criteria:

* women with Brest Cancer undergoing adjutant Radiation therapy

Exclusion Criteria:

* previous history of RT, MRM,
* concomitant presence of two or more malignant tumors
* metastasis to other areas
* allergy or intolerance to tahini
* skin diseases and wounds
* severe liver and renal disease
* autoimmune diseases
* pregnant and lactating women
* those who treated with hypo fraction RT

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-08 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
severity of dermatitis | 4 weeks
  Change from Baseline severity at 4 weeks. The radiation dermatitis will be assessed according to the Radiation Therapy Oncology Group/ European Organization for Research and Treatment of Cancer (RTOG/EORTC) scales